CLINICAL TRIAL: NCT01320748
Title: fMRI Study of a Dual Process Treatment Protocol With Substance Dependent Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inova Health Care Services (Other)
Collaborators: George Mason University (Other); Georgetown University (Other)
Responsible Party: Principal Investigator, Maria Hadjiyane, Senior Director Behavioral Health Adult Ambulatory Services, Inova Health Care Services
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IHS 11-001
Record Dates: First submitted 2011-03-07; First posted 2011-03-22 (Estimated); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Substance Abuse; Substance Dependence; Alcohol Abuse; Drug Use; Relapse
Keywords: Abstinence from alcohol; Substance Abuse and Mental Health Services; Social Support; Psychosocial Support Systems; Psychological support; Cognitive Support; Emotional Support; Mental Support; Psychosocial Support; Intervention Studies; Prevention & control; Preventive therapy; Treatment; Therapy; Magnetic Resonance Imaging; fMRI; Imaging; Magnetic Resonance Imaging, Functional; MRI Scans; MRI, Functional; Clinical Protocols; Protocols, Treatment; Drug Abuse Treatment Center; Substance Abuse Treatment Center
MeSH Terms: conditions — Substance-Related Disorders; Alcoholism; Recurrence | interventions — Psychotherapy, Group; Secondary Prevention

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dual Processing (Experimental)
  Interventions: Behavioral: Dual Processing
- Relapse Prevention (Active Comparator)
  Interventions: Behavioral: Relapse Prevention

INTERVENTIONS:
Behavioral: Dual Processing — A 10-week, 20-session program, which meets two times per week for 2 hours each time. It is a psychosocial intervention that combines a visual processing (structured drawing activities to engage in sensory-based cue exposure) and a verbal processing component (structured cognitive-behavioral therapy). The treatment focuses on sensory-based emotional expression and cognitive reappraisal and containment strategies that facilitate emotional regulation around a patient's drug and alcohol use experiences.
  Other Names: Group Therapy; DP
  Arms: Dual Processing
Behavioral: Relapse Prevention — The program's standard care outpatient program is a Relapse Prevention 10-week, 20-session, psychosocial intervention program, which meets two times per week for 2 hours each time. This RP program is based on Gorski's Relapse Prevention model and is a primarily didactic approach.
  Other Names: Group Therapy; RP
  Arms: Relapse Prevention

SUMMARY:
The purpose of this study is to determine whether drug-dependent adults who participate in a dual processing relapse prevention treatment protocol that allows for sensory-based exposure experiences over 10-weeks in outpatient treatment will show significant brain change related to diminished cue reactivity, and greater improvement in self-efficacy, anxiety, somatization, and treatment retention, as compared to the standard care patients in a relapse prevention program.

DETAILED DESCRIPTION:
The substance abuse literature consistently shows that negative emotional states and subjective stress are highly predictive of relapse and significantly influence behavioral motivation. From a neurobiological perspective, stress associated with withdrawal and substance abuse experiences stimulates chemical and hormonal changes in the brain creating a protracted hyperaroused state. Further, cognitive control resources (i.e., cognitive coping skills/relapse prevention training) have been shown to exert minimal impact on behavioral decision-making in the presence of intense affective material. Thus, implicit cognitive processes play a significant role in drug use behavior, decreasing self regulation capacities and increasing risk of. Specifically, high levels of stress can compromise prefrontal cortex functioning, with the nucleus accumbens, orbitofrontal cortex and amygdala functional changes related to increased cue reactivity.

Taken together, the current literature strongly suggests that verbally-based therapies may have limited utility as a singular form of treatment in early substance abuse recovery, as the brain may not be functionally ready for executive level processing. Instead, the multidisciplinary substance abuse literature suggests that psychosocial treatment methods need to include a range of learning approaches that allow for visual-sensory processing, in addition to traditional verbal-based processing. Integrated multi-modal interventions are needed to offer opportunities for activation of these different brain regions to facilitate cognitive-affective balance in behavioral decision-making.

ELIGIBILITY:
Study Inclusion Criteria:

* Age < 18 years old
* Signed informed consent for this study
* History of chemical dependency
* Meets Inova CATS Relapse Prevention admission criteria
* Must have at least 60 days of sobriety prior to admission with documentation of negative drug and alcohol screening
* Documentation of HIV negative test result (completed in the past year)
* Willing and able to attend an out-patient drug treatment group for two hours twice a week for 10 weeks
* Willing to complete study-required evaluations (including assessments, questionnaires, drug/alcohol testing, week 8 qualitative interview)
* A score < 25 on the MoCA (Montreal Cognitive Assessment)

Study Exclusion Criteria:

* History of taking "anti-craving" medication in the past 90 days
* Other medical illness or florid psychiatric symptoms that would render the participant inappropriate for study participation
* History of receiving treatment for addictions other than substance use (i.e. food, gambling, sex)
* Clinical determination of dementia or organic brain syndrome
* History of major head injury
* Incapable of consenting for themselves due to cognitive impairment
* Enrollment in another study that might interfere with analysis of this study

Additional Inclusion Criteria for fMRI sub-study:

* Willing and able to participate in the fMRI arm of the study
* If of childbearing capacity, must have negative screening urine pregnancy test and be willing to use birth control as specified in the consent document

Additional Exclusion Criteria for fMRI sub-study:

* Left-handed
* Cardiac pacemakers or other body metals
* Other criteria identified on the "MRI Screening Form" that would indicate that having an MRI would be unsafe
* Pregnancy
* Claustrophobia (for the fMRI testing)
* Muscular or back problems that would prevent participant from being able to lie in the scanner for 90 minutes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2011-02; Primary Completion 2012-03 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
fMRI blood-oxygenation-level-dependent (BOLD) signal change as a measure of emotional reactivity related to the visual presentation of drug-imagery. | 10 weeks
  In a subset of approximately 26 subjects, fMRI technology will be employed to examine brain structure and function change (pre-treatment and post-treatment) in the amygdaloid region, orbitofrontal cortex, in the anterior cingluate cortex (structure implicated in drug cue attention); in medial prefrontal cortex and right dorsolateral prefrontal cortex (associated with effective behavioral decision-making in substance abusers).

SECONDARY OUTCOMES:
Heart rate during MRI scanning as a measure of emotional reactivity related to the visual presentation of drug-imagery. | 10 weeks
  Changes in heart rate related to the visual presentation of drug-imagery during MRI scanning, to assess cue reactivity differences across the treatment and control groups at two time-points (pre-intervention and post-intervention).
Quality of Life Inventory (QOLI) as a measure of the subject's quality of life. | 10 weeks
  Questionnaire completed by subjects at baseline and at the end of the study. We will measure changes in Overall QOLI score and Weighted Satisfaction Profile score at the two time-points (pre-intervention and post-intervention).
Brief Symptoms Inventory (BSI), as a measure of subjective craving, anxiety, and somatization | 10 weeks
  Questionnaire completed by subjects at baseline and at the end of the study. We will measure changes in Nonpatient T Score and Percentile in the 12 domains at the two time-points (pre-intervention and post-intervention).
Hamilton - Depression Inventory (HAM-D) as a measure of depression. | 10 weeks
  Questionnaire completed by subjects at baseline and at the end of the study. We will measure changes in the total Hamilton depression scale score at the two time-points (pre-intervention and post-intervention).
Urine specimen toxicology analysis as a measure of treatment retention. | Weekly for 10 weeks
  Urine specimen collection and analysis to track patient drug use on a weekly basis during the 10 weeks in treatment.
Blood Alcohol Level analysis as a measure of treatment retention. | Weekly for 10 weeks
  Breathalizer test for alcohol to track patient alcohol use on a weekly basis during the 10 weeks in treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Holly C Matto, PhD, Principal Investigator — Virginia Commonwealth University, School of Social Work
Locations (2):
- United States (2):
  - Georgetown Center for Functional And Molecular Imaging, Georgetown University Medical Center, Washington D.C., District of Columbia
  - Inova Heath Services Comprehensive Addictions Treatment Services (ICATS), Falls Church, Virginia

REFERENCES:
- [Background] Brewer JA, Potenza MN. The neurobiology and genetics of impulse control disorders: relationships to drug addictions. Biochem Pharmacol. 2008 Jan 1;75(1):63-75. doi: 10.1016/j.bcp.2007.06.043. Epub 2007 Jul 3. PMID 17719013
- [Background] Brewin CR. A cognitive neuroscience account of posttraumatic stress disorder and its treatment. Behav Res Ther. 2001 Apr;39(4):373-93. doi: 10.1016/s0005-7967(00)00087-5. PMID 11280338
- [Background] Brewin CR, Dalgleish T, Joseph S. A dual representation theory of posttraumatic stress disorder. Psychol Rev. 1996 Oct;103(4):670-86. doi: 10.1037/0033-295x.103.4.670. PMID 8888651
- [Background] Charney DS. Psychobiological mechanisms of resilience and vulnerability: implications for successful adaptation to extreme stress. Am J Psychiatry. 2004 Feb;161(2):195-216. doi: 10.1176/appi.ajp.161.2.195. PMID 14754765
- [Background] Chee MW, Sriram N, Soon CS, Lee KM. Dorsolateral prefrontal cortex and the implicit association of concepts and attributes. Neuroreport. 2000 Jan 17;11(1):135-40. doi: 10.1097/00001756-200001170-00027. PMID 10683845
- [Background] Childress AR, Ehrman RN, Wang Z, Li Y, Sciortino N, Hakun J, Jens W, Suh J, Listerud J, Marquez K, Franklin T, Langleben D, Detre J, O'Brien CP. Prelude to passion: limbic activation by "unseen" drug and sexual cues. PLoS One. 2008 Jan 30;3(1):e1506. doi: 10.1371/journal.pone.0001506. PMID 18231593
- [Background] Coffey SF, Stasiewicz PR, Hughes PM, Brimo ML. Trauma-focused imaginal exposure for individuals with comorbid posttraumatic stress disorder and alcohol dependence: revealing mechanisms of alcohol craving in a cue reactivity paradigm. Psychol Addict Behav. 2006 Dec;20(4):425-35. doi: 10.1037/0893-164X.20.4.425. PMID 17176177
- [Background] Fein G, Di Sclafani V, Meyerhoff DJ. Prefrontal cortical volume reduction associated with frontal cortex function deficit in 6-week abstinent crack-cocaine dependent men. Drug Alcohol Depend. 2002 Sep 1;68(1):87-93. doi: 10.1016/s0376-8716(02)00110-2. PMID 12167554
- [Background] Goldin PR, McRae K, Ramel W, Gross JJ. The neural bases of emotion regulation: reappraisal and suppression of negative emotion. Biol Psychiatry. 2008 Mar 15;63(6):577-86. doi: 10.1016/j.biopsych.2007.05.031. Epub 2007 Sep 21. PMID 17888411
- [Background] Goldstein M, Brendel G, Tuescher O, Pan H, Epstein J, Beutel M, Yang Y, Thomas K, Levy K, Silverman M, Clarkin J, Posner M, Kernberg O, Stern E, Silbersweig D. Neural substrates of the interaction of emotional stimulus processing and motor inhibitory control: an emotional linguistic go/no-go fMRI study. Neuroimage. 2007 Jul 1;36(3):1026-40. doi: 10.1016/j.neuroimage.2007.01.056. Epub 2007 Mar 12. PMID 17509899
- [Background] Goodman A. Neurobiology of addiction. An integrative review. Biochem Pharmacol. 2008 Jan 1;75(1):266-322. doi: 10.1016/j.bcp.2007.07.030. Epub 2007 Jul 27. PMID 17764663
- [Background] Houben K, Schoenmakers TM, Wiers RW. I didn't feel like drinking but I don't know why: the effects of evaluative conditioning on alcohol-related attitudes, craving and behavior. Addict Behav. 2010 Dec;35(12):1161-3. doi: 10.1016/j.addbeh.2010.08.012. Epub 2010 Aug 11. PMID 20810220
- [Background] Koob GF. The neurobiology of addiction: a neuroadaptational view relevant for diagnosis. Addiction. 2006 Sep;101 Suppl 1:23-30. doi: 10.1111/j.1360-0443.2006.01586.x. PMID 16930158
- [Background] Matto HC, Strolin-Goltzman J. Integrating social neuroscience and social work: innovations for advancing practice-based research. Soc Work. 2010 Apr;55(2):147-56. doi: 10.1093/sw/55.2.147. PMID 20408356
- [Background] Matto HC, Strolin JS, Mogro-Wilson C. A pilot study of a dual processing substance user treatment intervention with adults. Subst Use Misuse. 2008;43(3-4):285-94. doi: 10.1080/00952990701202848. PMID 18365931
- [Background] Matto H. A bio-behavioral model of addiction treatment: applying dual representation theory to craving management and relapse prevention. Subst Use Misuse. 2005;40(4):529-41. doi: 10.1081/ja-200030707. PMID 15830734
- [Background] Moeller SJ, Maloney T, Parvaz MA, Dunning JP, Alia-Klein N, Woicik PA, Hajcak G, Telang F, Wang GJ, Volkow ND, Goldstein RZ. Enhanced choice for viewing cocaine pictures in cocaine addiction. Biol Psychiatry. 2009 Jul 15;66(2):169-76. doi: 10.1016/j.biopsych.2009.02.015. Epub 2009 Apr 9. PMID 19358975
- [Background] Ochsner KN, Ray RD, Cooper JC, Robertson ER, Chopra S, Gabrieli JD, Gross JJ. For better or for worse: neural systems supporting the cognitive down- and up-regulation of negative emotion. Neuroimage. 2004 Oct;23(2):483-99. doi: 10.1016/j.neuroimage.2004.06.030. PMID 15488398
- [Background] Phan KL, Wager T, Taylor SF, Liberzon I. Functional neuroanatomy of emotion: a meta-analysis of emotion activation studies in PET and fMRI. Neuroimage. 2002 Jun;16(2):331-48. doi: 10.1006/nimg.2002.1087. PMID 12030820
- [Background] Schneider F, Habel U, Wagner M, Franke P, Salloum JB, Shah NJ, Toni I, Sulzbach C, Honig K, Maier W, Gaebel W, Zilles K. Subcortical correlates of craving in recently abstinent alcoholic patients. Am J Psychiatry. 2001 Jul;158(7):1075-83. doi: 10.1176/appi.ajp.158.7.1075. PMID 11431229
- [Background] Shaham Y, Erb S, Stewart J. Stress-induced relapse to heroin and cocaine seeking in rats: a review. Brain Res Brain Res Rev. 2000 Aug;33(1):13-33. doi: 10.1016/s0165-0173(00)00024-2. PMID 10967352
- [Background] Tanabe J, Tregellas JR, Dalwani M, Thompson L, Owens E, Crowley T, Banich M. Medial orbitofrontal cortex gray matter is reduced in abstinent substance-dependent individuals. Biol Psychiatry. 2009 Jan 15;65(2):160-4. doi: 10.1016/j.biopsych.2008.07.030. Epub 2008 Sep 18. PMID 18801475
- [Background] Uhl GR, Drgon T, Johnson C, Fatusin OO, Liu QR, Contoreggi C, Li CY, Buck K, Crabbe J. "Higher order" addiction molecular genetics: convergent data from genome-wide association in humans and mice. Biochem Pharmacol. 2008 Jan 1;75(1):98-111. doi: 10.1016/j.bcp.2007.06.042. Epub 2007 Jul 25. PMID 17764662
- [Background] van Reekum CM, Johnstone T, Urry HL, Thurow ME, Schaefer HS, Alexander AL, Davidson RJ. Gaze fixations predict brain activation during the voluntary regulation of picture-induced negative affect. Neuroimage. 2007 Jul 1;36(3):1041-55. doi: 10.1016/j.neuroimage.2007.03.052. Epub 2007 Apr 6. PMID 17493834
- See also: Inova Health System, Comprehensive Addiction Treatment Services (CATS) — http://inova.org/cats
- See also: National Institute on Drug Abuse — http://www.nida.nih.gov/NIDAHome.html